CLINICAL TRIAL: NCT07041060
Title: Evaluation of the Efficacy and Safety of a Nutraceutical Containing Sodium Alginate, Sodium Bicarbonate, PEA, a Blend of Opuntia Ficus Indica, and Olea Europaea, Musa Paradisiaca, and Ginger in Patients With NERD
Brief Title: Evaluation of the Efficacy and Safety of Eolo in Patients With NERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Carlo Calabrese, Clinical Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DIMEC, University of Bologna
Record Dates: First submitted 2025-05-30; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Non-erosive Reflux Disease; Reflux Disease, Gastro-Esophageal; Nutraceutical
Keywords: non erosive reflux Disease; nutraceutical treatment
MeSH Terms: conditions — Non-Erosive Reflux Disease; Gastroesophageal Reflux | interventions — Proton Pump Inhibitors

STUDY DESIGN:
Intervention Model Description: Group A: Patients receiving Eolo + half-dose PPIs for 12 weeks, then Eolo alone for 12 additional weeks.
  Group B: Patients receiving half-dose PPIs alone for 12 weeks, then Eolo alone for 12 additional weeks.
  Group C: Patients receiving half-dose PPIs only for 24 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Active Comparator): half-dose PPIs for 24 weeks
  Interventions: Dietary Supplement: EOLO; Dietary Supplement: Group C: Eolo
- Group B (Experimental): Patients receiving half-dose PPIs alone for 12 weeks, then Eolo alone for 12 additional weeks.
  Interventions: Drug: PPI (proton pump inhibitor); Dietary Supplement: Group C: Eolo
- Group A (Experimental): Patients receiving Eolo 24 we
  Interventions: Drug: PPI (proton pump inhibitor)

INTERVENTIONS:
Dietary Supplement: EOLO — Eolo, a nutraceutical blend of sodium alginate, sodium bicarbonate, palmitoylethanolamide (PEA), and herbal extracts
  Arms: Group C
Drug: PPI (proton pump inhibitor) — Received a half-dose of PPIs for 24 weeks
  Arms: Group A; Group B
Dietary Supplement: Group C: Eolo — Eolo, a nutraceutical blend of sodium alginate, sodium bicarbonate, palmitoylethanolamide (PEA), and herbal extracts for 24 weeks
  Arms: Group B; Group C

SUMMARY:
Background: Non-erosive reflux disease (NERD) is a prevalent subtype of gastroesophageal reflux disease (GERD), often inadequately managed with proton pump inhibitors (PPIs) alone. Eolo, a nutraceutical blend of sodium alginate, sodium bicarbonate, palmitoylethanolamide (PEA), and herbal extracts, has been proposed as an adjunctive therapy to enhance symptom relief and mucosal protection.

Objective: This study evaluates the efficacy and safety of a nutraceutical [Eolo®, Cristalfarma s.r.l. - Milan (IT)] in combination with PPIs or alone compared to PPIs therapy in patients with NERD.

Methods: A single-center, randomized, parallel-group study was conducted, enrolling 60 patients with NERD. Participants were randomized into three groups: (A) Eolo + half-dose PPIs for 12 weeks, (B) half-dose PPIs alone for 12 weeks, and (C) a control group receiving only half-dose PPIs for 24 weeks. After 12 weeks, groups A and B discontinued PPIs and continued with Eolo alone for an additional 12 weeks. Symptom relief and quality of life (QoL) were assessed using GERD-HRQOL and RSI questionnaires at baseline (T0), 12 weeks (T1), and 24 weeks (T2).

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of a nutraceutical in combination with PPIs or alone compared to PPIs therapy in patients with NERD.

A single-center, randomized, parallel-group study was conducted, enrolling 60 patients with NERD. Participants were randomized into three groups: (A) Eolo + half-dose PPIs for 12 weeks, (B) half-dose PPIs alone for 12 weeks, and (C) a control group receiving only half-dose PPIs for 24 weeks. After 12 weeks, groups A and B discontinued PPIs and continued with Eolo alone for an additional 12 weeks. Symptom relief and quality of life (QoL) were assessed using GERD-HRQOL and RSI questionnaires at baseline (T0), 12 weeks (T1), and 24 weeks (T2).

ELIGIBILITY:
Inclusion Criteria:Participants were eligible for the study if they met the following criteria:

* Had a diagnosis of non-erosive reflux disease (NERD) with typical reflux symptoms persisting for at least three months and occurring at least three times per week in the month preceding the study screening visit.
* Were aged between 18 and 80 years.
* Had been on therapy with a proton pump inhibitor (PPI) at a standard dosage for at least six weeks (40 mg pantoprazole/esomeprazole, 30 mg lansoprazole, or 20 mg omeprazole/rabeprazole).
* Had a diagnosis of NERD confirmed by the absence of macroscopic lesions of the distal esophageal mucosa on endoscopy performed within six months before the screening visit and a positive score on a validated questionnaire (Reflux Disease Questionnaire, RDQ Score ≥ 8).

Exclusion Criteria:Patients were excluded if they had any of the following conditions:

* Erosive esophagitis or Barrett's esophagus.
* Gastric or duodenal ulcer.
* History of major gastric or gastrointestinal surgery.
* Atopy or food intolerances.
* Thyroid disease.
* Diabetes or metabolic syndrome.
* Pregnancy or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Symptom relief and quality of life (QoL) | Baseline (T0), Week 12 (T1), and Week 24 (T2). Score range 0-50; higher scores indicate worse quality of life.
  GERD-HRQOL

SECONDARY OUTCOMES:
RSI (Reflux Symptom Index) | Baseline (T0), Week 12 (T1), and Week 24 (T2). Score range 0-45; higher scores indicate worse symptoms.
  Reflux Symptom Index

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Calabrese, Prof of Gastroenterology, PI, Principal Investigator — University of Bologna
Locations (1):
- DIMEC, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code